CLINICAL TRIAL: NCT03102944
Title: Minicare BNP Normal Value Study - MI-BNP-CE02-NV2016
Brief Title: Determining Normal Values of BNP Levels for the Minicare BNP IVD Assay.
Status: Completed | Type: Observational
Sponsor: Philips Handheld Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: HHDx-07998
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Leftover plasma samples (without cells/ RNA/DNA) will be aliquoted and stored at Sponsor for potential future analysis/ projects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy volunteers: no intervention, extra blood tube taken with blood donation at bloodbank and blood is tested on IVD away from patient.
  Interventions: Diagnostic Test: Minicare BNP

INTERVENTIONS:
Diagnostic Test: Minicare BNP — no real intervention since only leftover materials are used from volunteers and samples are not tested on Minicare BNP IVD device near any volunteer.

SUMMARY:
Main objective is to determine normal values for Brain Natriuretic Peptide (BNP) levels for the Minicare BNP using K2-EDTA (ethylenediaminetetraacetic acid ) venous whole blood and K2-EDTA plasma samples from healthy subjects.

K2-EDTA whole blood and K2-EDTA plasma samples from approximately 150 normal healthy volunteer, preferably 50% men and 50% women, will be analysed using the Minicare BNP system. This will be a single-center study. The study will consist of a 1-day visit for each study subject on which screening based on a questionnaire, blood draw and discharge will occur. For each eligible subject, K2-EDTA whole blood will be collected and both K2-EDTA whole blood and K2-EDTA plasma will be analyzed using the Minicare BNP. Blood donors, presenting voluntarily at one of the Sanquin posts in, the Netherlands (e.g Eindhoven) will be checked on health status and selected based on 2 questionnaires. The collected K2-EDTA whole blood tubes from eligible subjects will be transferred from the Sanquin posts to Philips Eindhoven for Minicare BNP testing. From one subject, both K2-EDTA whole blood and K2-EDTA plasma will be measured in singleton. K2-EDTA whole blood and plasma will be measured within 6 hours after blood collection. The data obtained will be used for determination of normal values of BNP in a healthy population. Leftover plasma samples (without cells/ RNA/DNA) will be aliquoted and stored at Philips for potential future analysis/ projects). Testing will be done according to a DRAFT Instructions for use (IFU) of the Minicare BNP.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Willing and able to sign the informed consent form (ICF)

Exclusion Criteria:

* Subjects suffering from cardiac and/or vascular disease, renal dysfunction, hypertension, cancer, Chronic Obstructive Pulmonary Disease (COPD), instable diabetes, pregnancy and extreme overweight are not allowed to donate blood.
* Subjects with a history of cardiac and/or vascular disease, renal dysfunction, cancer, COPD or instable diabetes are not allowed to donate blood.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
Normal values for BNP for the Minicare BNP | 4 weeks
  To determine normal values for BNP levels for the Minicare BNP using K2- EDTA venous whole blood and K2-EDTA plasma samples from healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Diederick Keizer, Study Chair — Clinical Affairs Manager
Locations (1):
- Philips EB Handheld Diagnostics, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: No